CLINICAL TRIAL: NCT06833905
Title: Combining Virtual Reality and Hypnosis to Alleviate Chronic Pain in Elderly Patients with Hand Arthritis: a Pilot Randomized Clinical Trial
Brief Title: Combining Virtual Reality and Hypnosis to Alleviate Chronic Pain in Elderly Patients with Hand Arthritis
Acronym: VRHArthrisis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-3539
Record Dates: First submitted 2025-01-13; First posted 2025-02-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Arthritis; Arthritis/Arthrosis; Arthritis, Rheumatoid; Elderly
Keywords: virtual reality; hypnosis; arthritis; pain; quality of life; elderly
MeSH Terms: conditions — Arthritis; Osteoarthritis; Arthritis, Rheumatoid; Pain

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined virtual reality and hypnosis (Experimental): The intervention consist in 4 different sessions with the VR headset, two consisting in presenting landscapes (i.e., beach, forest) and two consisting in hypnosis techniques (i.e., magic hand, manipulating hand).
  Interventions: Behavioral: Virtual reality: Beach; Behavioral: Virtual Reality: Forest; Behavioral: Hypnosis: Magic Hand; Behavioral: Hypnosis: Pain Manipulation; Behavioral: Session 1bis - 1 week; Behavioral: Follow-up
- Waiting list (No Intervention): The control group consist in a waiting list.

INTERVENTIONS:
Behavioral: Virtual reality: Beach — Session 1 or 2 (counterbalanced): Exposure to a beach landscape
  Arms: Combined virtual reality and hypnosis
Behavioral: Virtual Reality: Forest — Session 1 or 2 (counterbalanced): Exposure to a forest landscape
  Arms: Combined virtual reality and hypnosis
Behavioral: Hypnosis: Magic Hand — Session 3 or 4 (counterbalanced): Exposure to a hypnosis technique: the magic hand
  Arms: Combined virtual reality and hypnosis
Behavioral: Hypnosis: Pain Manipulation — Session 3 or 4 (counterbalanced): Exposure to a hypnosis technique: manipulating the pain
  Arms: Combined virtual reality and hypnosis
Behavioral: Session 1bis - 1 week — Repetition of the Session 1 one week after Session 4
  Arms: Combined virtual reality and hypnosis
Behavioral: Follow-up — Repetition of the Session 1 three weeks after Session 4
  Arms: Combined virtual reality and hypnosis

SUMMARY:
The goal of this pilot randomized clinical trial is to test the efficacy of an intervention combining virtual reality and hypnosis on decreasing pain and improving quality of life in elderly patients with hand arthritis. The main questions it aims to answer are:

* Does the intervention allow for an improvement of patient reported outcomes related to pain and quality of life?
* Does the intervention allow for an improvement of physiological variables related to pain? Researchers will compare intervention group to a passive control group (i.e., waiting list with treatment as usual).

Participants in the intervention group will be provided a virtual reality headset allowing them to beneficiate from the virtual reality and hypnosis modules.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in French
* Being diagnosed with hand arthrisis
* Reporting an invalidating chronic pain in hand related to the condition

Exclusion Criteria:

* Experiencing a medical condition altering the ability to consent or participate in the study
* Experiencing cognitive disorders; Experiencing sensory disorders (deafness, blindness)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Perceived pain | Intervention group: Two times per week (before and after each session)/Control group: One time per week, For all: from enrollment to the end of intervention at 6 weeks and at a 3 weeks follow-up
  Brief Pain Inventory - Short Form (BPI-SF) ; 9 items ; Scores from 0 to 10 ; scores are computed into mean score ; higher scores mean higher levels of pain (negative outcome)

SECONDARY OUTCOMES:
Anxiodepressive symptoms | Intervention group: Two times per week (before and after each session)/Control group: One time per week, For all: from enrollment to the end of intervention at 6 weeks and at a 3 weeks follow-up
  Hospital Anxiety and Depression Scale (HADS) ; 14 items: 7 items for anxiety, 7 items for depression ; Lickert scale from 0 to 3 ; a mean score is computed for each subscale (anxiety, depression) ; Minimum score for each scale: 0 ; Maximum score for each scale: 21 ; Higher scores mean worst symptomatology (negative outcome)
Quality of life | Intervention group: Two times per week (before and after each session)/Control group: One time per week, For all: from enrollment to the end of intervention at 6 weeks and at a 3 weeks follow-up
  Short-Form Health Survey 12 items (SF-12) ; includes 12 items measuring 8 dimensions (physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health) ; the physical (PCS-12) and mental (MCS-12) scales are transformed to have a mean of 50 and a standard deviation of 10 in the general U.S. population ; participants' scores represent the difference compared to the population average (measured in standard deviations) ; scores above 50 indicate a better-than-average health-related quality of life (positive outcome), while scores below 50 suggest below-average health-related quality of life (negative outcome).
Fatigue | From enrollment, each week during 6 weeks, Intervention group: Two times per week (before and after each session)
  Multidimensional Fatigue Inventory - 10 Items (MFI-10) ; 10 items measuring 5 dimensions (general fatigue, physical fatigue, mental fatigue, reduction in activity and reduction in motivation) ; the Lickert scale ranges from 1 to 5 ; the answer on the scale represents the score of each individual item which is then added up to a sum for each dimension ; scores per dimension can vary between 4 and 20 ; higher scores indicate higher fatigue levels (negative outcome)
Relaxation | From enrollment, each week during 6 weeks, Intervention group: Two times per week (before and after each session)
  Relaxation State Questionnaire (RSQ) ; 10 items ; Lickert scales from 1 to 5 ; scores are computed into a mean score; higher scores indicate higher levels of relaxation (positive outcome)
Perceived changes | From Session 2, each week during 5 weeks, Intervention group: Two times per week (before and after each session)
  Three free items evaluating perceived change in pain, anxiodepressive symptoms, and quality of life ; Lickert scale ranging from 1 to 10 ; higher scores indicate greater perceived changes (positive outcome)
Cybersickness | From enrollment, each week during 6 weeks, Intervention group: One time per week (after each session)
  Cybersickness questionnaire ; 16 items including 2 subscales (nausea and oculomotor); Lickert scale ranging from 0 to 3 ; scores for each subscale are summed to give final scores ; higher scores indicate higher levels of cybersickness (negative outcome)

OTHER OUTCOMES:
Respiratory frequence | One time per week, from enrollment to the end of treatment at 6 weeks, during the whole hypnosis session (for Intervention group) or during 15 minutes where the subject is not engaging in any task (for Control group)
  Will be calculated with the XDCF module in BIOPAC MP200-WS (Biopac Systems, Goleta, CA) ; A higher respiratory frequence is a negative outcome as it indicates higher levels of anxiety and lower levels of relaxation.
Heart rate | One time per week, from enrollment to the end of treatment at 6 weeks, during the whole hypnosis session (for Intervention group) or during 15 minutes where the subject is not engaging in any task (for Control group)
  Will be calculated with module RSP & ECG Bionomadix (Amplificator RPEC-R) in BIOPAC MP200-WS (Biopac Systems, Goleta, CA) ; A higher heart rate is a negative outcome as it indicates higher levels of anxiety and lower levels of relaxation
Electrodermal activity | One time per week, from enrollment to the end of treatment at 6 weeks, during the whole hypnosis session (for Intervention group) or during 15 minutes where the subject is not engaging in any task (for Control group)
  Will be calculated with module EDA Bionomadix in BIOPAC MP200-WS (Biopac Systems, Goleta, CA) ; A higher electrodermal activity is a negative outcome as it indicates higher levels of anxiety and lower levels of relaxation
Heart rate variability | One time per week, from enrollment to the end of treatment at 6 weeks, during the whole hypnosis session (for Intervention group) or during 15 minutes where the subject is not engaging in any task (for Control group)
  Will be calculated with module EDA Bionomadix in BIOPAC MP200-WS (Biopac Systems, Goleta, CA) ; A higher heart rate variability is a positive outcome as it indicates lower levels of anxiety and higher levels of relaxation
Prescribed treatment with level 1 or 2 analgesics (self-reported) | The measure will be taken at 3 timepoints: once at enrollment, once at Week 4, and once during the Follow-up session 9 weeks after the enrollment
  Daily frequency intake of prescribed analgesics reported by the patient
Prescribed treatment with level 1 or 2 analgesics (medical record) | The measure will be taken at 3 timepoints: once at enrollment, once at Week 4, and once during the Follow-up session 9 weeks after the enrollment
  Daily frequency intake of prescribed analgesics reported by the patient's medical record (dose written on their prescription)
Prescribed treatment with level 1 or 2 anxiolytics (self-reported) | The measure will be taken at 3 timepoints: once at enrollment, once at Week 4, and once during the Follow-up session 9 weeks after the enrollment
  Daily frequency intake of prescribed anxiolytics reported by the patient
Patient demand for medical prescription | The measure will be taken at 3 timepoints: once at enrollment, once at Week 4, and once during the Follow-up session 9 weeks after the enrollment
  Patient demand for medical prescription (requested dose/intake frequency) retrieved in medical record
Clinical consultations for pain | The measure will be taken at 3 timepoints: once at enrollment, once at Week 4, and once during the Follow-up session 9 weeks after the enrollment
  Frequency of clinical consultations for pain
Prescribed treatment with level 1 or 2 antidepressants (medical record) | The measure will be taken at 3 timepoints: once at enrollment, once at Week 4, and once during the Follow-up session 9 weeks after the enrollment
  Daily frequency intake of prescribed antidepressants reported by the patient's medical record (dose written on their prescription)
Prescribed treatment with level 1 or 2 antidepressants (self-reported) | The measure will be taken at 3 timepoints: once at enrollment, once at Week 4, and once during the Follow-up session 9 weeks after the enrollment
  Daily frequency intake of prescribed antidepressants reported by the patient
Prescribed treatment with level 1 or 2 anxiolytics (medical record) | The measure will be taken at 3 timepoints: once at enrollment, once at Week 4, and once during the Follow-up session 9 weeks after the enrollment
  Daily frequency intake of prescribed anxiolytics reported by the patient's medical record (dose written on their prescription)

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared in a dedicated OSF repository.
Supporting Information: Study Protocol, SAP
Time Frame: Supporting information will be available from the definitive publication of results.
Access Criteria: All IPD that underlie results in a publication will be shared in a dedicated OSF repository.

REFERENCES:
- [Derived] Fournier V, Simard MF, Yuen SY, Guine J, Rousseaux F, Lebeau J, Jerbi K, Richebe P, Landry M, Rainville P, Ogez D. Combining virtual reality and hypnosis to alleviate chronic pain in elderly with hand arthritis: protocol for a randomised phase II clinical trial. BMJ Open. 2025 Oct 5;15(10):e103841. doi: 10.1136/bmjopen-2025-103841. PMID 41047257